CLINICAL TRIAL: NCT06905548
Title: A Critical Intervention for Sustainable Health: Climate Change Awareness of Executive Nurses: a Randomized Controlled Trial
Brief Title: Climate Change Awareness: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Collaborators: Maltepe University (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst. Prof., University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Climate Change Awareness
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthcare Professionals; Sustainability; Climate Change
Keywords: randomized controlled trial; sustainable healthcare; educational intervention; climate change awareness; Nurse managers

STUDY DESIGN:
Intervention Model Description: This study employs a randomized controlled trial (RCT) design to assess the impact of an educational intervention on nurse managers' awareness of climate change and its implications for healthcare. Participants will be randomly assigned to either an intervention group receiving structured climate change and healthcare sustainability training or a control group receiving no intervention. The training includes theoretical and interactive sessions on climate-related health risks, mitigation strategies, and sustainable hospital practices. Baseline and post-intervention data will be collected using validated instruments, including the Climate Change Awareness Scale. The study aims to determine whether targeted education can enhance climate change awareness among nurse managers and support environmentally responsible decision-making in healthcare settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group: Climate Change Awareness Education (for the group receiving the training) (Experimental): (for the group receiving the training)
  Interventions: Behavioral: climate change awareness training
- Control Group: No Educational Intervention (No Intervention): (for the group that does not receive the training)

INTERVENTIONS:
Behavioral: climate change awareness training — The climate change training planned for nurse managers consists of 4 sessions of 2 days, each lasting 40 minutes.
  Arms: Intervention Group: Climate Change Awareness Education (for the group receiving the training)

SUMMARY:
Background: Climate change awareness among nurse managers is crucial for enhancing healthcare efficiency and mitigating environmental and societal impacts. This study aims to develop and implement an educational program to improve nurse managers' awareness of climate change.

Methods: A randomized controlled trial will be conducted with 108 nurse managers (54 experimental, 54 control) from two major hospitals in Istanbul, Turkey: Kartal Dr. Lütfi Kırdar City Hospital (n=71) and Göztepe Prof. Dr. Süleyman Yalçın City Hospital (n=58). Sample size was determined using G*Power 3.1.9.7, referencing the study by Alvarez-Nieto et al. (2022), assuming an effect size of 0.79, a significance level of α=0.05, and 95% power. The required sample size was calculated as 90, increased by 20% to account for potential attrition, resulting in 108 participants.

Participants will be recruited through full enumeration sampling due to the limited number of nurse managers. Data will be collected via face-to-face administration of a Demographic Information Form (12 items) and the Climate Change Awareness Scale (Ataklı & Kuran, 2022), which consists of 52 items rated on a 5-point Likert scale, with a reliability coefficient (α) of 0.92.

Intervention: Following institutional approval from the Provincial Health Directorate, education nurses will disseminate information about the study via digital communication platforms. Nurse managers will be enrolled in separate digital groups for experimental and control conditions. Pre-test data will be collected face-to-face before the intervention. The educational program will be delivered to the experimental group, while the control group will receive no intervention. Post-test data collection will occur four weeks after the intervention.

Statistical Analysis: Nominal and ordinal data will be presented as frequencies and percentages, while scale scores will be reported as means and standard deviations or medians and ranges. Normality of data distribution will be assessed using the Kolmogorov-Smirnov test. Independent Samples T-Test and One-Way ANOVA will be used for normally distributed variables, while Mann-Whitney U and Kruskal-Wallis tests will be used for non-normally distributed data. Analyses will be conducted using SPSS 26 with a significance level set at p<0.05.

Expected Outcomes: The study will evaluate the effectiveness of the educational program in enhancing climate change awareness among nurse managers. Findings will contribute to the development of targeted training programs to integrate environmental awareness into nursing leadership.

Ethical Considerations: Ethical approval and institutional permissions will be obtained prior to study commencement.

DETAILED DESCRIPTION:
Background and Rationale: Climate change poses significant challenges to public health and healthcare systems. Nurse managers play a crucial role in implementing environmentally sustainable healthcare practices and mitigating the negative effects of climate change on health services. Despite the increasing awareness of climate change among healthcare professionals, structured educational programs aimed at enhancing nurse managers' knowledge and attitudes regarding this issue are needed. This study aims to evaluate the effectiveness of an educational intervention in improving nurse managers' awareness of climate change.

Study Objectives: This study's primary objective is to assess an educational program's impact on nurse managers' awareness of climate change. Specific objectives include:

Measuring the baseline level of climate change awareness among nurse managers. Evaluating the effectiveness of the educational intervention in enhancing their awareness.

Identifying factors associated with higher awareness levels.

Methods:

Study Design:

A randomized controlled trial (RCT) will be conducted with a pre-test and post-test design.

Study Setting and Population:

The study will be conducted at two major hospitals: Kartal Dr. Lütfi Kırdar City Hospital and Göztepe Prof. Dr. Süleyman Yalçın City Hospital. The target population consists of nurse managers working in these hospitals.

Sample Size Calculation: The study aims to include 108 nurse managers, with 54 in the experimental and 54 in the control groups. Sample size calculation was performed using G*Power 3.1.9.7 based on the effect size reported in the study by Alvarez-Nieto et al. (2022). An effect size of 0.79 (d = 0.79), 5% significance level (α = 0.05), and 95% power (1-β = 0.95) were used to determine a required sample size of 90 participants. To account for potential dropouts, the sample size was increased by 20%, resulting in a final target of 108 participants.

Sampling Method:

A census sampling method will be used to include all eligible nurse managers in the study setting. Since the number of nurse managers is limited, this method ensures maximum representation.

Intervention: The educational intervention will include a structured training program on climate change awareness. The program will include:

The science of climate change and its health implications. The role of healthcare professionals in mitigating climate change. Strategies for implementing sustainable practices in healthcare settings. The training will be delivered via interactive workshops and online modules over a four-week period.

Data Collection Tools:

Data will be collected through:

Demographic Information Form: A 12-item questionnaire covering age, gender, education level, work experience, and prior climate change training.

Climate Change Awareness Scale: Developed by Ataklı and Kuran (2022), this 52-item, five-factor Likert scale measures climate change awareness, issue perception, knowledge of causes, concerns, and expected policies. Higher scores indicate greater awareness. The scale has a Cronbach's alpha reliability coefficient of 0.92.

Data Collection Process:

Institutional approvals will be obtained from the Provincial Health Directorate.

The study will be introduced to nurse managers via hospital education nurses, who will disseminate information and collect voluntary participation lists.

Participants will be randomized into experimental and control groups. Pre-test data will be collected before the intervention. The educational program will be delivered to the experimental group. Four weeks after the intervention, post-test data will be collected from both groups.

Data Analysis:

Descriptive statistics (frequency, percentage, mean, standard deviation) will summarize demographic and baseline characteristics.

The normality of scale scores will be assessed using the Kolmogorov-Smirnov test.

Independent samples t-test will be used for normally distributed continuous variables.

Mann-Whitney U test will be applied for non-normally distributed variables. One-way ANOVA or the Kruskal-Wallis test will be used for comparisons across multiple groups.

All statistical analyses will be conducted using SPSS 26.0 with a significance level of p < 0.05.

Ethical Considerations: The study will adhere to ethical principles, including obtaining informed consent from participants. Institutional Review Board (IRB) approval will be obtained before data collection.

Expected Outcomes: The study is expected to demonstrate that a structured educational program significantly improves nurse managers' awareness of climate change. The findings will contribute to developing sustainable healthcare policies and training programs tailored to healthcare leaders.

Conclusion: Addressing climate change awareness among nurse managers is essential for sustainable healthcare delivery. This study's results will provide evidence-based recommendations for integrating climate change education into nursing leadership programs.

ELIGIBILITY:
Inclusion Criteria:

* Nurse managers working in Kartal Dr. Lütfi Kırdar City Hospital and Göztepe Prof. Dr. Süleyman Yalçın City Hospital.
* Individuals who have at least one year of managerial experience in a healthcare setting.
* Participants who voluntarily agree to participate in the study and provide informed consent.
* Individuals who can complete both pre-test and post-test assessments.

Exclusion Criteria:

* Nurse managers who are currently on leave (e.g., maternity, sick leave).
* Individuals who have participated in a similar educational program on climate change awareness in the past year.
* Those who do not consent to participate in the study.
* Participants who fail to complete the required assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Climate Change Awareness Score Time Frame | 4 months
  Baseline and 4 weeks post-intervention Description: The difference in scores obtained from the Climate Change Awareness Scale before and after the educational program. Higher scores indicate indicate increased awareness.

IPD SHARING:
Plan to Share IPD: No